CLINICAL TRIAL: NCT02048631
Title: Retrospective Analysis Of Sensory Recovery Of Donor Size And Related Quality Life In Oral Cancer Patients Receiving Free Flap Reconstruction
Brief Title: Analysis Of Sensory Recovery Of Donor Size And Quality Life In Oral Cancer Patients
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB-20130085
Record Dates: First submitted 2013-10-08; First posted 2014-01-29 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2013-07

CONDITIONS: Oral Cancer
Keywords: oral cancer,Quality of life,Sensory
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Oral Cancer Patients underwent Free Flap Reconstruction

SUMMARY:
The aim of the study is to investigate post-surgery sensory impairment and life quality changes in oral cancer patients who underwent free flap (Free Flap) on post-operative 6 months, 12 months, and 24 months, respectively

ELIGIBILITY:
Inclusion Criteria:

1. patients with American Society of Anesthesiologists physical status I-III
2. Older than 20 patients
3. Diagnosis of oral canaer ,requiring free flap reconstruction

Exclusion Criteria:

1. Diagnosis of a serious mental illness involving formal thought disorder (e.g., schizophrenia) documented in medical record
2. Cognitive with dementia, delirium

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Oral Cancer Patients Receiving Free Flap Reconstruction
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
sensory impairment on Donor site | up to 2 years
  comparison the contra-lateral side and donor site; measurement of thermal hyperalgesia with thermal roller temperatures measurement of allodynia with brush and cotton swab measurment of mechanical hyperalgesia with Von Frey filaments sensory impairments with roller wheel

SECONDARY OUTCOMES:
postoperative life quality using EORTC QLQ C-30 questionnaire . | postoperative 6 months to one year, postoperative 1 to 2 years, and over postoperative 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kao Pin Chang, MD,PhD., Study Director — Department of Plastic Surgery,Kaohsiung Medical University,Taiwan
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan